CLINICAL TRIAL: NCT05788861
Title: French Pediatric Nationwide Observatory of Invasive Group A Streptococcal Infection (in Childen for 0 to 18 Ages)
Brief Title: Invasive Group A Streptococcal Infection
Acronym: ISAI
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Other Study IDs: ISAI
Record Dates: First submitted 2022-12-22; First posted 2023-03-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Sepsis Due to Streptococcus, Group A; Risk Factors; Severe Infection; Medical Care; Medical Complications; Outcome, Fatal; Therapy; Strain; Virulence Factors
MeSH Terms: conditions — Infections; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is observational, retrospective and prospective study in pediatric patients hospitalized with invasive streptococcal A infection

DETAILED DESCRIPTION:
The main of this study is to identify and record cases of invasive and severe infections due to Streptococcus pyogenes. In order to evaluate the incidence of severe forms of disease and the possible contributing factors, and to optimize their management.

Admitted patients to intensive care or critical care units in reported via Santé Publique France may also be included in this study.

Secondly, epidemiological, clinical, bacteriological data of all severe or not cases, of group A Streptococcal infections will be compiled to describe their characteristics, and try to explain this recrudescence as well as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age<18 years
* Documented invasive Group A Streptococcus infection (identification of GAS in a normally sterile site or from another site in case of toxin shock or necrotizing dermo-hypodermatitis)

Exclusion Criteria:

* Opposition of the patient or his/her legal representative

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatrics patients with documented invasive infection due to Group A Streptococcus
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalisation | 1 year
  How long patient was hospitalised during this infection
Treatments provided in intensive care unit | 1 year
  what treatments are used in intensive care unit to treat infection
Complications | 1 year
  what are the complications due to severe infection
Treatments used in routine care unit | 1 year
  which treatments are used in routine care unit to treat the infection
Risk factors | 1 year
  description of underlying conditions
Characterization of Group A Streptococcus strains | 1 year
  Characterization of Group A Streptococcus strains by the CNR
Death | 1 year
  Death Outcome during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Yves Gillet, Principal Investigator — hôpital Femme-Mère-Enfant, Bron; Camille Brehin, Principal Investigator — HOPITAUX MERE et ENFANTS CHU TOULOUSE; Lionel Berthomieu, Principal Investigator — University Hospital, Toulouse; Corinne Levy, Study Director — Association Clinique Thérapeutique Infantile du val de Marne
Locations (1):
- ACTIV, Créteil, France